CLINICAL TRIAL: NCT00505219
Title: Multi-center Clinical Trial of the Application of Ixmyelocel-T in the Treatment of Osteonecrosis of the Femoral Head
Brief Title: Ixmyelocel-T Treatment of Patients With Osteonecrosis of the Femoral Head
Acronym: ON-CORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABI 55-0705-1
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Osteonecrosis
Keywords: Osteonecrosis
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ixmyelocel-T (Experimental): Core decompression & treatment with Tissue Repair Cells (TRCs), demineralized bone matrix bound in autologous plasma
  Interventions: Biological: Ixmyelocel-T
- Standard of Care Only (Active Comparator): Core decompression, demineralized bone matrix bound in autologous plasma, without any TRCs.
  Interventions: Other: Standard of Care Only

INTERVENTIONS:
Biological: Ixmyelocel-T — Core decompression of the femoral head to remove necrotic tissue with Ixmyelocel-T given to treatment arm only.
  Arms: Ixmyelocel-T
Other: Standard of Care Only — Core decompression of the femoral head to remove necrotic tissue
  Arms: Standard of Care Only

SUMMARY:
The purpose of this study is to determine if Ixmyelocel-T grafting with demineralized bone matrix bound in autologous plasma after core decompression surgery is superior to core decompression with demineralized bone matrix bound in autologous plasma in preventing progression of osteonecrosis to a more severe disease stage (Stage II to III or higher) from the time of surgery until 24 months later, in patients with University of Pennsylvania (UPenn) Stage IIB or C disease at diagnosis.

DETAILED DESCRIPTION:
This study is an event-driven, multi-center, prospective, independent observer-blinded, controlled, randomized Phase III clinical trial enrolling patients diagnosed with University of Pennsylvania (Steinberg) Classification Stage IIB or C osteonecrosis of the femoral head.

* The first patient group is the Treatment Group and will receive core decompression and treatment with BRCs and demineralized bone matrix bound in autologous plasma, and
* The second patient group is the Control Group and will receive core decompression and demineralized bone matrix bound in autologous plasma, without any BRCs.
* Enrollment: With an anticipated drop-out rate of 10% in up to twenty (20) sites, a total of approximately 135 patients will be enrolled and randomized to obtain 120 evaluable patients (75 for the TRC treatment group and 45 for the Control treatment group).
* Primary endpoint: The percentage of patients progressing to a more severe UPenn disease stage (Stage II to III or higher) between 0 and 24 months will be the primary efficacy variable to demonstrate TRC therapy is superior to Control therapy.

ELIGIBILITY:
Inclusion Criteria:

* UPenn (Steinberg) classification of osteonecrosis, inclusive of Stages IIB and IIC. Diagnosis will be based on magnetic resonance imaging (MRI).
* Modified index of necrotic extent < 40
* Idiopathic and non-idiopathic osteonecrosis.
* No infection in affected bones at the time of surgery.
* Patient competent to give informed consent.
* Normal organ and marrow function defined as:

  * Leukocytes ≥ 3000/µL;
  * Absolute neutrophil count ≥ 1500/µL;
  * Platelets ≥ 140,000/µL;
  * Serum AST (SGOT)/ALT (SGPT) < 2.5 X institutional standard range;
  * Serum creatinine within normal limits, based on clinical laboratory normal range.
* Female patients not pregnant or lactating.
* Patients with a history of corticosteroids or on active therapy, will only be eligible for enrollment if corticosteroid use is suspended for 1 month prior and 6 months after cell therapy and surgery.
* Patients who have been treated with oral bisphosphonates are eligible for the trial if treatment was stopped at least 6 months prior to enrollment.

Exclusion Criteria:

* Stages IA, IB, IC, IIA, IIIA or more severe femoral head osteonecrosis, primarily based on diagnosis by MRI.
* Flattening of the femur head (UPenn Stage IV) or articular cartilage collapse at the time of core decompression surgery.
* Septic arthritis; stress fracture, or non-osteonecrosis metabolic bone diseases (e.g., Paget's disease of bone, osteogenesis imperfecta, primary hyperparathyroidism, fibrous dysplasia [monostotic, polyostotic McCune-Albright syndrome] and osteopetrosis).
* Any active bisphosphonate treatment or any history of intravenous (IV) treatment
* HIV, syphilis, positive at time of screening.
* Active hepatitis B or hepatitis C infection at the time of screening
* Known allergies to protein products (horse or bovine serum, or porcine trypsin).
* Patients who will require continuous, systemic, high dose corticosteroid therapy (more than 7.5 mg/day) within 6 months after surgery.
* Patients in active treatment for cancer or blood dyscrasia, or have received chemotherapy, radiotherapy or immunotherapy in the past 2 years.
* Immunodeficiency diseases.
* Participation in another clinical study in the past 30 days or concurrent participation in another clinical trial.
* History of regular alcohol consumption exceeding 2 drinks/day (1 drink = 5 oz [150 mL] of wine or 12 oz [360 mL] of beer or 1.5 oz [45 mL] of hard liquor) within 6 months of screening and/or history of illicit drug use.
* MRI-incompatible internal devices (pacemakers, aneurysm clips, etc)
* Body mass index (BMI) of 40 Kg/m2 or greater
* Patients unable to tolerate general anesthesia defined as an American Society of Anesthesiologists (ASA) criteria of > 2
* Patients with poorly controlled diabetes mellitus (HbA1C > 8%), or with peripheral neuropathy, or known concomitant vascular problems.
* Patients receiving treatment with hematopoietic growth factors or anti-vasculogenesis or anti-angiogenesis treatment
* Traumatic osteonecrosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The progression of patients with UPenn Stage IIB or IIC disease to a more severe stage based on all available x-ray and MRI imaging. Patients who have a definitive procedure but do not have a valid assessment will be considered to have progressed. | 24 months

SECONDARY OUTCOMES:
Time to progression (in months) | 24 months
Osteonecrosis volume measured by MRI | 24 months
Pain and quality of life questionnaires | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Hungerford, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - University of Minnesota Department of Orthopaedic Surgery, Minneapolis, Minnesota
  - Lutheran Medical Center, Brooklyn, New York